CLINICAL TRIAL: NCT04066920
Title: Clinical Efficacy and Safety of IBER Salvage Treatment Followed by Ibrutinib Maintenance for Transplant-ineligible Patients With Relapsed or Refractory Primary Central Nervous System Lymphoma (PCNSL): a Multicenter, Single-arm, Prospective Phase II Study
Brief Title: IBER Salvage Treatment Followed by Ibrutinib Maintenance for Relapsed or Refractory PCNSL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Deok-Hwan Yang (Other)
Responsible Party: Sponsor-Investigator, Deok-Hwan Yang, Professor, Chonnam National University Hospital
Organization: Chonnam National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBER
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Primary Central Nervous System Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBER treatment arm (Experimental): This is the only arm in a single-arm phase II study.
  Interventions: Drug: IBER salvage chemotherapy followed by ibrutinib maintenance therapy

INTERVENTIONS:
Drug: IBER salvage chemotherapy followed by ibrutinib maintenance therapy — Induction therapy with IBER (up to 6 cycles) [ Ibrutinib 560 mg/d on D1-21 + Rituximab 375 mg/m2 on D1 (on D1/8/15 in C1) + Ifosfamide 3.75 g/m2 on D2 + Etoposide 100 mg/m2 on D2-4 ], followed by ibrutinib 560 mg/d maintenance therapy for up to 6 months

SUMMARY:
This is a multicenter, single-arm, prospective phase II study to evaluate the efficacy and safety of a novel combination regimen for relapsed/refractory PCNSL. Specifically, ibrutinib will be administered in combination with ifosfamide, etoposide and rituximab (IBER) as a salvage chemotherapy, which is followed by maintenance ibrutinib monotherapy of fixed duration.

DETAILED DESCRIPTION:
Given the limited activity of salvage therapy with high-dose methotrexate re-treatment and/or alkylator-based treatment in patients with relapse or refractory PCNSL, the development of novel salvage chemotherapy regimen remains an area of clinical unmet need.

Ibrutinib, an oral inhibitor of bruton tyrosine kinase (BTK), is known to induce death of diffuse large B-cell lymphoma (DLBCL) cells with dysregulated B-cell receptor (BCR) signaling and has shown promising activity in patients with a variety of B-cell malignancies. Recently, several studies reported that ibrutinib may have an excellent single-agent clinical activity against relapsed or refractory PCNSL. Furthermore, proven pharmacokinetic data suggested that ibrutinib successfully penetrated the BBB and reached the achievable concentration in cerebrospinal fluid. When ibrutinib is administered in combination with BBB-destructing chemotherapeutic agents (such as, temozolomide or etoposide) for salvage treatment of PCNSL, therefore, anti-lymphoma activity of ibrutinib could be maximized.

In this context, this phase II study is designed to evaluate the efficacy and safety of IBER salvage chemotherapy followed by ibrutinib maintenance for transplant ineligible patients with relapsed or refractory PCNSL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed PCNSL of CD20+ diffuse large B cell lymphoma (DLBCL)
* PCNSL relapsed or refractory after frontline methotrexate-based chemotherapy (with or without radiation therapy)
* At least one measurable lesion, which is defined as longest diameter of lesion > 0.5 cm, by contrast-enhanced MRI
* ECOG performance status 0-2
* Normal function of major organs

Exclusion Criteria:

* PCNSL other than DLBCL
* Primary ocular lymphoma
* PCNSL accompanied by systemic involvement
* Active infection with hepatitis B or C virus
* Known history of human immunodeficiency virus (HIV) infection
* Therapy with myelosuppressive chemotherapy or biologic therapy < 21 days prior to registration

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | From date of starting the study treatment until the date of finishing the study treatment for any reason, assessed up to 10 months
  The percentage of patients with a complete response (CR) or a partial response (PR)

SECONDARY OUTCOMES:
Safety and tolerability of the study treatment | From the first day of the first cycle of IBER induction chemotherapy to 30 days after the last dose of study drug, assessed up to 12 months
  Treatment-emergent adverse events graded according to the NCI-CTCAC version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Deok-Hwan Yang, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do, South Korea

REFERENCES:
- [Background] Villano JL, Koshy M, Shaikh H, Dolecek TA, McCarthy BJ. Age, gender, and racial differences in incidence and survival in primary CNS lymphoma. Br J Cancer. 2011 Oct 25;105(9):1414-8. doi: 10.1038/bjc.2011.357. Epub 2011 Sep 13. PMID 21915121
- [Background] Ferreri AJ, Abrey LE, Blay JY, Borisch B, Hochman J, Neuwelt EA, Yahalom J, Zucca E, Cavalli F, Armitage J, Batchelor T. Summary statement on primary central nervous system lymphomas from the Eighth International Conference on Malignant Lymphoma, Lugano, Switzerland, June 12 to 15, 2002. J Clin Oncol. 2003 Jun 15;21(12):2407-14. doi: 10.1200/JCO.2003.01.135. PMID 12805341
- [Background] Reni M, Mazza E, Foppoli M, Ferreri AJ. Primary central nervous system lymphomas: salvage treatment after failure to high-dose methotrexate. Cancer Lett. 2007 Dec 18;258(2):165-70. doi: 10.1016/j.canlet.2007.10.009. Epub 2007 Nov 13. PMID 17993246
- [Background] Fischer L, Thiel E, Klasen HA, Birkmann J, Jahnke K, Martus P, Korfel A. Prospective trial on topotecan salvage therapy in primary CNS lymphoma. Ann Oncol. 2006 Jul;17(7):1141-5. doi: 10.1093/annonc/mdl070. Epub 2006 Apr 7. PMID 16603598
- [Background] Reni M, Zaja F, Mason W, Perry J, Mazza E, Spina M, Bordonaro R, Ilariucci F, Faedi M, Corazzelli G, Manno P, Franceschi E, Pace A, Candela M, Abbadessa A, Stelitano C, Latte G, Ferreri AJ. Temozolomide as salvage treatment in primary brain lymphomas. Br J Cancer. 2007 Mar 26;96(6):864-7. doi: 10.1038/sj.bjc.6603660. Epub 2007 Feb 27. PMID 17325700
- [Background] Wilson WH, Young RM, Schmitz R, Yang Y, Pittaluga S, Wright G, Lih CJ, Williams PM, Shaffer AL, Gerecitano J, de Vos S, Goy A, Kenkre VP, Barr PM, Blum KA, Shustov A, Advani R, Fowler NH, Vose JM, Elstrom RL, Habermann TM, Barrientos JC, McGreivy J, Fardis M, Chang BY, Clow F, Munneke B, Moussa D, Beaupre DM, Staudt LM. Targeting B cell receptor signaling with ibrutinib in diffuse large B cell lymphoma. Nat Med. 2015 Aug;21(8):922-6. doi: 10.1038/nm.3884. Epub 2015 Jul 20. PMID 26193343
- [Background] Vater I, Montesinos-Rongen M, Schlesner M, Haake A, Purschke F, Sprute R, Mettenmeyer N, Nazzal I, Nagel I, Gutwein J, Richter J, Buchhalter I, Russell RB, Wiestler OD, Eils R, Deckert M, Siebert R. The mutational pattern of primary lymphoma of the central nervous system determined by whole-exome sequencing. Leukemia. 2015 Mar;29(3):677-85. doi: 10.1038/leu.2014.264. Epub 2014 Sep 5. PMID 25189415
- [Background] Braggio E, McPhail ER, Macon W, Lopes MB, Schiff D, Law M, Fink S, Sprau D, Giannini C, Dogan A, Fonseca R, O'Neill BP. Primary central nervous system lymphomas: a validation study of array-based comparative genomic hybridization in formalin-fixed paraffin-embedded tumor specimens. Clin Cancer Res. 2011 Jul 1;17(13):4245-53. doi: 10.1158/1078-0432.CCR-11-0395. Epub 2011 May 11. PMID 21562036
- [Background] Davis RE, Ngo VN, Lenz G, Tolar P, Young RM, Romesser PB, Kohlhammer H, Lamy L, Zhao H, Yang Y, Xu W, Shaffer AL, Wright G, Xiao W, Powell J, Jiang JK, Thomas CJ, Rosenwald A, Ott G, Muller-Hermelink HK, Gascoyne RD, Connors JM, Johnson NA, Rimsza LM, Campo E, Jaffe ES, Wilson WH, Delabie J, Smeland EB, Fisher RI, Braziel RM, Tubbs RR, Cook JR, Weisenburger DD, Chan WC, Pierce SK, Staudt LM. Chronic active B-cell-receptor signalling in diffuse large B-cell lymphoma. Nature. 2010 Jan 7;463(7277):88-92. doi: 10.1038/nature08638. PMID 20054396
- [Background] Grommes C, Pastore A, Palaskas N, Tang SS, Campos C, Schartz D, Codega P, Nichol D, Clark O, Hsieh WY, Rohle D, Rosenblum M, Viale A, Tabar VS, Brennan CW, Gavrilovic IT, Kaley TJ, Nolan CP, Omuro A, Pentsova E, Thomas AA, Tsyvkin E, Noy A, Palomba ML, Hamlin P, Sauter CS, Moskowitz CH, Wolfe J, Dogan A, Won M, Glass J, Peak S, Lallana EC, Hatzoglou V, Reiner AS, Gutin PH, Huse JT, Panageas KS, Graeber TG, Schultz N, DeAngelis LM, Mellinghoff IK. Ibrutinib Unmasks Critical Role of Bruton Tyrosine Kinase in Primary CNS Lymphoma. Cancer Discov. 2017 Sep;7(9):1018-1029. doi: 10.1158/2159-8290.CD-17-0613. Epub 2017 Jun 15. PMID 28619981
- [Background] Lionakis MS, Dunleavy K, Roschewski M, Widemann BC, Butman JA, Schmitz R, Yang Y, Cole DE, Melani C, Higham CS, Desai JV, Ceribelli M, Chen L, Thomas CJ, Little RF, Gea-Banacloche J, Bhaumik S, Stetler-Stevenson M, Pittaluga S, Jaffe ES, Heiss J, Lucas N, Steinberg SM, Staudt LM, Wilson WH. Inhibition of B Cell Receptor Signaling by Ibrutinib in Primary CNS Lymphoma. Cancer Cell. 2017 Jun 12;31(6):833-843.e5. doi: 10.1016/j.ccell.2017.04.012. Epub 2017 May 25. PMID 28552327
- [Background] Batchelor TT, Grossman SA, Mikkelsen T, Ye X, Desideri S, Lesser GJ. Rituximab monotherapy for patients with recurrent primary CNS lymphoma. Neurology. 2011 Mar 8;76(10):929-30. doi: 10.1212/WNL.0b013e31820f2d94. No abstract available. PMID 21383331
- [Background] Mappa S, Marturano E, Licata G, Frezzato M, Frungillo N, Ilariucci F, Stelitano C, Ferrari A, Soraru M, Vianello F, Baldini L, Proserpio I, Foppoli M, Assanelli A, Reni M, Caligaris-Cappio F, Ferreri AJ. Salvage chemoimmunotherapy with rituximab, ifosfamide and etoposide (R-IE regimen) in patients with primary CNS lymphoma relapsed or refractory to high-dose methotrexate-based chemotherapy. Hematol Oncol. 2013 Sep;31(3):143-50. doi: 10.1002/hon.2037. Epub 2012 Nov 14. PMID 23161567
- [Background] Birnbaum T, Stadler EA, von Baumgarten L, Straube A. Rituximab significantly improves complete response rate in patients with primary CNS lymphoma. J Neurooncol. 2012 Sep;109(2):285-91. doi: 10.1007/s11060-012-0891-7. Epub 2012 May 9. PMID 22570142
- [Background] Arellano-Rodrigo E, Lopez-Guillermo A, Bessell EM, Nomdedeu B, Montserrat E, Graus F. Salvage treatment with etoposide (VP-16), ifosfamide and cytarabine (Ara-C) for patients with recurrent primary central nervous system lymphoma. Eur J Haematol. 2003 Apr;70(4):219-24. doi: 10.1034/j.1600-0609.2003.00045.x. PMID 12656744
- [Background] Kuker W, Nagele T, Thiel E, Weller M, Herrlinger U. Primary central nervous system lymphomas (PCNSL): MRI response criteria revised. Neurology. 2005 Oct 11;65(7):1129-31. doi: 10.1212/01.wnl.0000178894.51436.54. PMID 16217075